CLINICAL TRIAL: NCT01425294
Title: A Multicenter, Non-interventional, Prospective Study to Collect Efficacy and Safety Data in Chinese Patients Who Have Received Faslodex 250mg Treatment Under the Condition of Actual Usage in Clinical Practice
Brief Title: Collection of Efficacy and Safety Data of Chinese Patients Who Have Received Faslodex 250mg Treatment
Status: Terminated | Type: Observational
Why Stopped: The study has been decided to be early terminated for the FAS 500 mg has launched in 2015. The use mothod of 250mg per month in clinical practice is off-label.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OCN-FAS-2011/1
Record Dates: First submitted 2011-08-19; First posted 2011-08-30 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: Chinese post-menopausal women; oestrogen receptor-positive locally advanced; metastatic breast cancer; fulvestrant 250 mg; failure to adjuvant anti-oestrogen therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is a post-authorisation study, committed to Center for Drug Evaluation (CDE) and China Food and Drug Administration (CFDA), in order to provide more effectiveness and safety data about Faslodex in real world clinical practice in China. The primary objective of this study was to evaluate the effectiveness of Faslodex 250mg monthly to treat post-menopausal women with oestrogen receptor-positive locally advanced or metastatic breast cancer, for disease relapse on or after adjuvant anti-oestrogen therapy or disease progression on therapy with an anti-oestrogen, in terms of progression-free survival (PFS), by collecting real world data according to Chinese physicians' clinical practice.

DETAILED DESCRIPTION:
A Multicenter, non-interventional, prospective study to collect effectiveness and safety data in Chinese patients who have received Faslodex treatment under the condition of actual usage in clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Chinese postmenopausal women with estrogen receptor positive, locally advanced or metastatic breast cancer Failure to previous anti-estrogen therapy, already received Faslodex 250mg treatment as determined by treating physician.
* The prescription of the Faslodex is clearly separated from the decision to include the subject in the NIS, and is part of normal medical practice. The recruitment of the patient to the study should be within 1 month of the first Faslodex injection.
* Provision of subject informed consent.

Exclusion Criteria:

* If participating in any controlled clinical trial, the subject cannot take part in this study.
* Hypersensitivity to the active substance, or to any of the other excipients.
* Pregnancy and lactation, or severe hepatic impairment.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical units
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2016-01-30 (Actual); Study Completion 2016-01-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of Faslodex 250mg monthly to treat post-menopausal women with ER+ locally advanced or MBC in terms of progression-free survival (PFS), by collecting real world data according to Chinese physicians' clinical practice. | Follow-up will be taken every 3 months after commencement of the protocol, through study completion, an average of 12 months.
  The primary objective of this study was to evaluate the effectiveness of Faslodex 250mg monthly to treat post-menopausal women with oestrogen receptor-positive locally advanced or metastatic breast cancer, for disease relapse on or after adjuvant anti-oestrogen therapy or disease progression on therapy with an anti-oestrogen, in terms of progression-free survival (PFS), by collecting real world data according to Chinese physicians' clinical practice.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Follow-up will be taken every 3 months after commencement of the protocol, through the study completion, an average of 12 months.
  ORR was defined as the percentage of patients who had a best objective tumour response of either complete response (CR) or partial response (PR) among the evaluable patients with measurable disease at baseline. The best overall response was the best response recorded from the start of the treatment until disease progression. The RECIST1.1 criteria were used to assess objective tumour response. ORR was summarized and expressed as the percentage together with the corresponding 95% confidence intervals (CI).
Frequency of Adverse Events | Follow-up will be taken every 3 months after commencement of the protocol, through study completion, an average of 12 months.
  Adverse events (AEs) data were coded using Medical dictionary for Regulatory Activities (MedDRA) version 14.0 and summarized by preferred term (PT) and system organ class (SOC).
Severity of Adverse Events | Follow-up will be taken every 3 months after commencement of the protocol, through study completion, an average of 12 months.
  SAEs causally related to study drug, AEs leading to discontinuation, AEs leading to death, respectively. Separate listings were provided for AEs causally related to study drug, AEs leading to death, respectively. The severity of all adverse events was analyzed according to CTCAE grading.

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (23):
- China (23):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Fuzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Guiyang, Guizhou
  - Research Site, Tangshan, Hebei
  - Research Site, Harbin, Heilongjiang
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Hohhot, Inner Mongolia
  - Research Site, Kunshan, Jiangsu
  - Research Site, Nanjing, Jiangsu
  - Research Site, Nantong, Jiangsu
  - Research Site, Xuzhou, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Qingdao, Shandong
  - Research Site, Weifang, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Kunming, Yunnan
  - Research Site, Hanghzou, Zhejiang
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Zhoushan, Zhejiang

REFERENCES:
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Wakeling AE, Dukes M, Bowler J. A potent specific pure antiestrogen with clinical potential. Cancer Res. 1991 Aug 1;51(15):3867-73. PMID 1855205
- [Background] Kansra S, Yamagata S, Sneade L, Foster L, Ben-Jonathan N. Differential effects of estrogen receptor antagonists on pituitary lactotroph proliferation and prolactin release. Mol Cell Endocrinol. 2005 Jul 15;239(1-2):27-36. doi: 10.1016/j.mce.2005.04.008. PMID 15950373
- [Background] Beverage JN, Sissung TM, Sion AM, Danesi R, Figg WD. CYP2D6 polymorphisms and the impact on tamoxifen therapy. J Pharm Sci. 2007 Sep;96(9):2224-31. doi: 10.1002/jps.20892. PMID 17518364
- [Background] Gallo MA, Kaufman D. Antagonistic and agonistic effects of tamoxifen: significance in human cancer. Semin Oncol. 1997 Feb;24(1 Suppl 1):S1-71-S1-80. PMID 9045319
- [Background] Osborne CK, Coronado-Heinsohn EB, Hilsenbeck SG, McCue BL, Wakeling AE, McClelland RA, Manning DL, Nicholson RI. Comparison of the effects of a pure steroidal antiestrogen with those of tamoxifen in a model of human breast cancer. J Natl Cancer Inst. 1995 May 17;87(10):746-50. doi: 10.1093/jnci/87.10.746. PMID 7563152
- [Background] Howell A, DeFriend D, Robertson J, Blamey R, Walton P. Response to a specific antioestrogen (ICI 182780) in tamoxifen-resistant breast cancer. Lancet. 1995 Jan 7;345(8941):29-30. doi: 10.1016/s0140-6736(95)91156-1. PMID 7799704
- [Background] Howell A, DeFriend DJ, Robertson JF, Blamey RW, Anderson L, Anderson E, Sutcliffe FA, Walton P. Pharmacokinetics, pharmacological and anti-tumour effects of the specific anti-oestrogen ICI 182780 in women with advanced breast cancer. Br J Cancer. 1996 Jul;74(2):300-8. doi: 10.1038/bjc.1996.357. PMID 8688341
- [Background] Howell A, Robertson JF, Quaresma Albano J, Aschermannova A, Mauriac L, Kleeberg UR, Vergote I, Erikstein B, Webster A, Morris C. Fulvestrant, formerly ICI 182,780, is as effective as anastrozole in postmenopausal women with advanced breast cancer progressing after prior endocrine treatment. J Clin Oncol. 2002 Aug 15;20(16):3396-403. doi: 10.1200/JCO.2002.10.057. PMID 12177099
- [Background] Osborne CK, Pippen J, Jones SE, Parker LM, Ellis M, Come S, Gertler SZ, May JT, Burton G, Dimery I, Webster A, Morris C, Elledge R, Buzdar A. Double-blind, randomized trial comparing the efficacy and tolerability of fulvestrant versus anastrozole in postmenopausal women with advanced breast cancer progressing on prior endocrine therapy: results of a North American trial. J Clin Oncol. 2002 Aug 15;20(16):3386-95. doi: 10.1200/JCO.2002.10.058. PMID 12177098
- See also: NIS-OCN-FAS-2011-1StudyReportSynopsisfinal — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=979&filename=NIS-OCN-FAS-2011-1StudyReportSynopsisfinal.docx